CLINICAL TRIAL: NCT04341597
Title: Evaluation of Transperineal Ultrasound Technic for Diagnostic Shorted Cervical Length for Pregnant Women (2nd and 3rd Trimester) Compared to Endovaginal Technic (Gold Standard)
Acronym: ECHO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: PI2018_843_0037
Record Dates: First submitted 2020-03-06; First posted 2020-04-10 (Actual); Last update posted 2025-09-19 (Actual); Status verified 2025-09

CONDITIONS: Ultrasound; Transperineal
Keywords: endovaginal; ultrasound; transperineal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- transperineal sonographic cervix assessment (Experimental)
  Interventions: Other: cervical ultrasound
- endovaginal sonographic cervix assessment (Active Comparator)
  Interventions: Other: cervical ultrasound

INTERVENTIONS:
Other: cervical ultrasound — All volunteer patients for whom a cervical ultrasound is indicated will have with a first operator the performing the usual technic, and with a second operator performing the trans perineal technic without being aware of the first measurement.

SUMMARY:
Endovaginal ultrasound is currently the gold standard to diagnose a shorted cervical length and, by extension, assess the risk of preterm labor. The major inconvenient is that this is an invasive method of diagnosis that tends to be poorly accepted by some patients. This study aims to evaluate the accuracy of a noninvasive transperineal ultrasound cervical measurement in comparison to the endovaginal technic in 2nd and 3nd trimester pregnant women where a cervical ultrasound is indicated.

DETAILED DESCRIPTION:
The cervical length is a crucial part of the diagnostic of premature labor. The gold standard technic is the endovaginal ultrasound. This is a technic with good reproducibility and good precision. Some authors have found the transperineal technic to present the same characteristics, without being as invasive. The aim of the study was to compare the results of the less invasive technic to the current invasive gold standard in pregnant women who consult for contraction, or for whom cervical modification is suspected in order to determine whether the former could replace the latter.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women between 2nd and 3rd trimester consulting in obstetric emergency for whom a cervical ultrasound is indicated

Exclusion Criteria:

* minor patients
* mentally deficient persons

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 85 (Actual)
Dates: Start 2020-03-06 (Actual); Primary Completion 2020-09-30 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
difference of measurement of the uterine cervix | at day 0
  difference of measurement of the uterine cervix will be done by analysing the variation between the transperineal measurement and endovaginal evaluation of the uterine cervix. Length will be measured in millimetres

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Amiens, Amiens, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Krief D, Foulon A, Tondreau A, Diouf M, Sergent F, Gondry J, Chevreau J. Transperineal ultrasound in routine uterine cervix measurement. Arch Gynecol Obstet. 2023 Feb;307(2):387-393. doi: 10.1007/s00404-022-06521-4. Epub 2022 Mar 23. PMID 35318500